CLINICAL TRIAL: NCT03463395
Title: Efficacy of Reza Band for the Treatment of Laryngopharyngeal Reflux
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for this study has ended and we were unable to enroll any subjects
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, John Rhee, Professor and Chairman, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO30948
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Laryngopharyngeal Reflux
MeSH Terms: conditions — Laryngopharyngeal Reflux

STUDY DESIGN:
Intervention Model Description: Sixty patients ≥ 18 years of age presenting to the investigator's laryngology outpatient clinic with LPR, with an RFS ≥ 7 and an RSI ≥ 13, not on anticoagulants, able to tolerate an endoscopy and consent to participate in this research study will be included. One cohort (Group A) will receive standard care (n =30), the other (Group B) will receive standard care plus the Reza band (to be worn as recommended by the manufacturer; n = 30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (No Intervention): Group A will receive standard of care
- Reza band use (Experimental): Group B will receive standard care plus the Reza band (worn as recommended by the manufacturer)
  Interventions: Device: Reza band

INTERVENTIONS:
Device: Reza band — Reza band, a non-medication, non-surgical medical device designed to reduce symptoms of LPR has recently been approved by the FDA. It works by stopping the flow of gastric contents through the upper esophageal sphincter (UES) by increasing the internal pressure of the UES
  Arms: Reza band use

SUMMARY:
We hypothesize that tissue and salivary pepsin will resolve after 12 weeks use of Reza Band, but not following standard of care alone. Additionally, RFS, RSI and inflammatory cytokines (IL -1β, -6, and -8) will decrease to normative levels following 12 weeks use of Reza Band, but not with standard of care alone.

Primary Objective The primary objective is to evaluate the efficacy of the Reza Band for the treatment of LPR. We propose a pilot clinical trial to test the hypothesis that the Reza Band is effective for the treatment of LPR, measured by resolution of pepsin and decrease to normative values for RSI, Reflux Finding Score (RFS) and inflammatory cytokines.

The long-term goal is to determine the efficacy of the Reza Band in the sequential progression of reflux-attributed laryngeal inflammatory and neoplastic disease.

DETAILED DESCRIPTION:
We propose a prospective cohort study. Sixty patients ≥ 18 years of age presenting to our laryngology outpatient clinic with LPR, with an RFS ≥ 7 and an RSI ≥ 13, not on anticoagulants, able to tolerate an endoscopy and consent to participate in this research study will be included. The study will consist of two cohorts. Cohort one will receive standard care (n = 30), and cohort two will receive standard care plus the Reza Band (to be worn as recommended by the manufacturer; n = 30). Patients will be assigned to either of the cohorts, based on their preferences.

Two laryngeal (posterior cricoid) biopsy specimens (one for pepsin ELISA and the other for qPCR for IL -1β, -6, and -8 inflammatory cytokines) and a throat saliva sample (for pepsin ELISA) will be obtained pre- and posttreatment (12 weeks) in an ambulatory clinic setting. The RSI, a patient-reported symptom severity questionnaire, will be administered in the clinic pre- and posttreatment. (36) Patients will be instructed to cough and clear the back of their throat to provide a saliva sample prior to endoscopy. The RFS (37) will be obtained by the study physicians during office endoscopy prior to biopsy. Deidentified biopsy and saliva samples will be transported to the research laboratory on ice and stored at -80 prior to analyses by ELISA and qPCR.

Pepsin ELISA One biopsy per subject will be homogenized in urea lysis buffer and total protein concentration determined as previously described (28). Saliva samples will be cleared by brief centrifugation. Noncompetitive indirect sandwich enzyme-linked immunosorbent assay described previously (35) will be performed to detect pepsin in biopsy homogenate and saliva.

qPCR RNA will be extracted from a second biopsy, DNAsed and reverse transcribed as described (38). Real time polymerase chain reaction will be performed in a Viaa7 Real Time PCR System using Taqman Gene Expression Assays targeting IL -1β, -6, and -8, and the housekeeping gene HPRT1 (ThermoFisher Scientific, Waltham, MA).

This pilot study will pave the way for clinical trials of a much-needed therapy for airway reflux. If the hypothesis proves true and the Reza Band resolves pepsin and inflammatory cytokines, and significantly improves endoscopic signs (RFS) and symptoms (RSI) of LPR, these data will also support a clinical trial to assess the utility of the Reza Band in preventing reflux-attributed laryngeal inflammatory and neoplastic disease sequelae. To our knowledge, this is the first study that will use pepsin as a primary outcome measure; it is believed to be a sensitive and specific biomarker for reflux and aspiration.

Deidentified biopsy and saliva samples will be transported to the research laboratory on ice and stored at -80 degrees C prior to analyses by ELISA and qPCR. The tissue and saliva samples will be labeled with patient study ID number and date of collection.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of laryngopharyngeal reflux (LPR).
2. Age ≥ 18 years.
3. Reflux Finding Score (RFS) of ≥ 7 and an Reflux Symptom Index (RSI) ≥ 13.
4. Patients should be able to tolerate an endoscopy.
5. Patients must be deemed able to comply with the treatment plan and follow-up schedule.
6. Enrollment on an interventional postoperative study is allowed if study device/agents do not overlap i.e. no other investigational device or medication for the treatment of LPR is permitted during the duration of this study.
7. Patients must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

1. Patient should not be on anticoagulants
2. Currently being treated with another investigational medical device and/or drug.
3. Currently receiving treatment for sleep apnea with continuous positive airway pressure (CPAP).
4. The patient is female and is of childbearing potential and is not using an acceptable method of birth control or is pregnant or breast-feeding.
5. Previous head or neck surgery or radiation.
6. Carotid artery disease, thyroid disease or history of cerebral vascular disease.
7. Suspected esophageal cancer.
8. Has either a pacemaker or implanted cardioverter defibrillator (ICD).
9. Nasopharyngeal cancer.
10. Previously undergone Nissen Fundoplication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in Tissue and Salivary Pepsin Levels | The change in Pepsin will be measured pre and post 12 week treatment for LPR +/- Reza band
  The primary objective is to evaluate the efficacy of the Reza Band for the treatment of LPR. We propose a pilot clinical trial to test the hypothesis that the Reza Band is effective for the treatment of LPR, measured by resolution of pepsin and decrease to normative values for RSI, Reflux Finding Score (RFS) and inflammatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Nikki Johnston, PhD, Study Director — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
If the decision is made to make individual participant data (IPD) available to other researchers, that data will be completely identified prior to release.

REFERENCES:
- [Background] Ford CN. Evaluation and management of laryngopharyngeal reflux. JAMA. 2005 Sep 28;294(12):1534-40. doi: 10.1001/jama.294.12.1534. PMID 16189367
- [Background] Koufman JA. The otolaryngologic manifestations of gastroesophageal reflux disease (GERD): a clinical investigation of 225 patients using ambulatory 24-hour pH monitoring and an experimental investigation of the role of acid and pepsin in the development of laryngeal injury. Laryngoscope. 1991 Apr;101(4 Pt 2 Suppl 53):1-78. doi: 10.1002/lary.1991.101.s53.1. PMID 1895864
- [Background] Vaezi MF. Extraesophageal manifestations of gastroesophageal reflux disease. Clin Cornerstone. 2003;5(4):32-8; discussion 39-40. doi: 10.1016/s1098-3597(03)90097-4. PMID 15101493
- [Background] GABRIEL CE, JONES DG. The importance of chronic laryngitis. J Laryngol Otol. 1960 Jun;74:349-57. doi: 10.1017/s0022215100056693. No abstract available. PMID 13825824
- [Background] Yudkin PL, Aboualfa M, Eyre JA, Redman CW, Wilkinson AR. New birthweight and head circumference centiles for gestational ages 24 to 42 weeks. Early Hum Dev. 1987 Jan;15(1):45-52. doi: 10.1016/0378-3782(87)90099-5. PMID 3816638
- [Background] Perrier D, Gibaldi M. Clearance and biologic half-life as indices of intrinsic hepatic metabolism. J Pharmacol Exp Ther. 1974 Oct;191(1):17-24. No abstract available. PMID 4423599
- [Background] Inokuchi K. [Prospectives on cancer treatment in the future--from its clinical aspects]. Gan To Kagaku Ryoho. 1987 May;14(5 Pt 2):1372-9. Japanese. PMID 3109325
- [Background] Wight R, Paleri V, Arullendran P. Current theories for the development of nonsmoking and nondrinking laryngeal carcinoma. Curr Opin Otolaryngol Head Neck Surg. 2003 Apr;11(2):73-7. doi: 10.1097/00020840-200304000-00002. PMID 14515082
- [Background] Koufman JA. Low-acid diet for recalcitrant laryngopharyngeal reflux: therapeutic benefits and their implications. Ann Otol Rhinol Laryngol. 2011 May;120(5):281-7. doi: 10.1177/000348941112000501. PMID 21675582
- [Background] Koufman JA, Amin MR, Panetti M. Prevalence of reflux in 113 consecutive patients with laryngeal and voice disorders. Otolaryngol Head Neck Surg. 2000 Oct;123(4):385-8. doi: 10.1067/mhn.2000.109935. PMID 11020172
- [Background] Reulbach TR, Belafsky PC, Blalock PD, Koufman JA, Postma GN. Occult laryngeal pathology in a community-based cohort. Otolaryngol Head Neck Surg. 2001 Apr;124(4):448-50. doi: 10.1067/mhn.2001.114256. PMID 11283505
- [Background] Francis DO, Rymer JA, Slaughter JC, Choksi Y, Jiramongkolchai P, Ogbeide E, Tran C, Goutte M, Garrett CG, Hagaman D, Vaezi MF. High economic burden of caring for patients with suspected extraesophageal reflux. Am J Gastroenterol. 2013 Jun;108(6):905-11. doi: 10.1038/ajg.2013.69. Epub 2013 Apr 2. PMID 23545710
- [Background] Szczesniak MM, Williams RB, Brake HM, Maclean JC, Cole IE, Cook IJ. Upregulation of the esophago-UES relaxation response: a possible pathophysiological mechanism in suspected reflux laryngitis. Neurogastroenterol Motil. 2010 Apr;22(4):381-6, e89. doi: 10.1111/j.1365-2982.2009.01452.x. PMID 20377793
- [Background] Huszenicza G, Haraszti J, Molnar L, Solti L, Fekete S, Ekes K, Yaro AC. Some metabolic characteristics of dairy cows with different post partum ovarian function. Zentralbl Veterinarmed A. 1988 Aug;35(7):506-15. No abstract available. PMID 3142175
- [Background] Torrico S, Kern M, Aslam M, Narayanan S, Kannappan A, Ren J, Sui Z, Hofmann C, Shaker R. Upper esophageal sphincter function during gastroesophageal reflux events revisited. Am J Physiol Gastrointest Liver Physiol. 2000 Aug;279(2):G262-7. doi: 10.1152/ajpgi.2000.279.2.G262. PMID 10915633
- [Background] SELLICK BA. Cricoid pressure to control regurgitation of stomach contents during induction of anaesthesia. Lancet. 1961 Aug 19;2(7199):404-6. doi: 10.1016/s0140-6736(61)92485-0. No abstract available. PMID 13749923
- [Background] ANDERSEN N. Changes in intragastric pressure following the administration of suxamethonium. Preliminary report. Br J Anaesth. 1962 Jun;34:363-7. doi: 10.1093/bja/34.6.363. No abstract available. PMID 13861180
- [Background] Richards AJ, Walker SR, Paterson JW. A new anti-asthmatic drug (ICI 58 301): blood levels and spirometry. Br J Dis Chest. 1971 Oct;65(4):247-52. No abstract available. PMID 4332774
- [Background] Estler CJ, Ammon HP. Potentiation of the anticalorigenic action of the adrenergic beta-receptor antagonist MJ 1999 by cyclic 3',5'-AMP. Life Sci. 1969 Jul 1;8(13):759-64. doi: 10.1016/0024-3205(69)90266-5. No abstract available. PMID 4308507
- [Background] Lyon N, Gerlach J. Perseverative structuring of responses by schizophrenic and affective disorder patients. J Psychiatr Res. 1988;22(4):261-77. doi: 10.1016/0022-3956(88)90035-0. PMID 3216344
- [Background] Johnston N, Dettmar PW, Lively MO, Postma GN, Belafsky PC, Birchall M, Koufman JA. Effect of pepsin on laryngeal stress protein (Sep70, Sep53, and Hsp70) response: role in laryngopharyngeal reflux disease. Ann Otol Rhinol Laryngol. 2006 Jan;115(1):47-58. doi: 10.1177/000348940611500108. PMID 16466100
- [Background] Johnston N, Knight J, Dettmar PW, Lively MO, Koufman J. Pepsin and carbonic anhydrase isoenzyme III as diagnostic markers for laryngopharyngeal reflux disease. Laryngoscope. 2004 Dec;114(12):2129-34. doi: 10.1097/01.mlg.0000149445.07146.03. PMID 15564833
- [Background] Wassenaar E, Johnston N, Merati A, Montenovo M, Petersen R, Tatum R, Pellegrini C, Oelschlager B. Pepsin detection in patients with laryngopharyngeal reflux before and after fundoplication. Surg Endosc. 2011 Dec;25(12):3870-6. doi: 10.1007/s00464-011-1813-z. Epub 2011 Jun 22. PMID 21695583
- [Background] Hayat JO, Gabieta-Somnez S, Yazaki E, Kang JY, Woodcock A, Dettmar P, Mabary J, Knowles CH, Sifrim D. Pepsin in saliva for the diagnosis of gastro-oesophageal reflux disease. Gut. 2015 Mar;64(3):373-80. doi: 10.1136/gutjnl-2014-307049. Epub 2014 May 7. PMID 24812000
- [Background] Crapko M, Kerschner JE, Syring M, Johnston N. Role of extra-esophageal reflux in chronic otitis media with effusion. Laryngoscope. 2007 Aug;117(8):1419-23. doi: 10.1097/MLG.0b013e318064f177. PMID 17585281
- [Background] Knight J, Lively MO, Johnston N, Dettmar PW, Koufman JA. Sensitive pepsin immunoassay for detection of laryngopharyngeal reflux. Laryngoscope. 2005 Aug;115(8):1473-8. doi: 10.1097/01.mlg.0000172043.51871.d9. PMID 16094128
- [Background] Luebke K, Samuels TL, Chelius TH, Sulman CG, McCormick ME, Kerschner JE, Johnston N, Chun RH. Pepsin as a biomarker for laryngopharyngeal reflux in children with laryngomalacia. Laryngoscope. 2017 Oct;127(10):2413-2417. doi: 10.1002/lary.26537. Epub 2017 Feb 22. PMID 28224634
- [Background] Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice. 2002 Jun;16(2):274-7. doi: 10.1016/s0892-1997(02)00097-8. PMID 12150380
- [Background] Belafsky PC, Postma GN, Koufman JA. The validity and reliability of the reflux finding score (RFS). Laryngoscope. 2001 Aug;111(8):1313-7. doi: 10.1097/00005537-200108000-00001. PMID 11568561
- [Background] Samuels TL, Handler E, Syring ML, Pajewski NM, Blumin JH, Kerschner JE, Johnston N. Mucin gene expression in human laryngeal epithelia: effect of laryngopharyngeal reflux. Ann Otol Rhinol Laryngol. 2008 Sep;117(9):688-95. doi: 10.1177/000348940811700911. PMID 18834073